CLINICAL TRIAL: NCT03660228
Title: PTQA: A New Paradigm of Transfusion Decision Support for Patients With MDS
Brief Title: Peri-Transfusion QOL Assessments (PTQA): A New Paradigm of Transfusion Decision Support for Patients With MDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Vera and Joseph Dresner Foundation (Other)
Responsible Party: Principal Investigator, Gregory A. Abel, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-307
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-01

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS; Myelodysplastic Syndromes; Quality of life; Tranfusion-dependent
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peri-Transfusion QOL Assessment (Experimental): * Participants will be given a study packet containing a paper copy of the QUALMS
  * Study participants will fill out the survey on the day before their first/next pRBC transfusion.
  * Study participants will receive a second paper copy of the QUALMS, along with a stamped envelope addressed to the appropriate site
  * The second assessment will be scored and compared with the first, and both the patient and provider will be sent a report with the results
  Interventions: Other: Peri-Transfusion QOL Assessment

INTERVENTIONS:
Other: Peri-Transfusion QOL Assessment — Participants will undergo a peri-transfusion quality of life assessment (PTQA) using the Quality of Life in Myelodysplasia Scale (QUALMS)

SUMMARY:
This research study is evaluating how to best tailor blood transfusion decisions to match the quality of life changes experienced by individual patients with MDS.

DETAILED DESCRIPTION:
Each patient with MDS reacts differently to blood transfusions; some will feel better after transfusion, while others may not. The main purpose of this survey study is to determine whether it is possible to use quality of life changes - as measured by a validated questionnaire - experienced by individual patients to help physicians and patients with MDS make decisions regarding future blood transfusions. This research is being done because the investigators hope to help doctors better understand the impact of blood transfusions on the quality of life of each patient.

The study uses a standardized MDS-specific quality of life questionnaire that participants will fill out before and after an upcoming transfusion. The investigators will compare the scores of these questionnaires and notify both the participant and provider if the participant has experienced any changes (positive or negative) in his/her quality of life before and after transfusion. The investigators' hope is that doctor-patient teams will use this quality of life information to determine whether the participant should continue receiving transfusions, decrease the frequency of transfusions, or stop receiving transfusions altogether if not needed.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age
* Patients with MDS
* Patients approaching an Hb of 8.5 g/dL during enrollment period OR
* Patients with >1 transfusion scheduled during an 8-week period
* Ability to read and understand English

Exclusion Criteria:

* Age <18 years
* Cr > 2
* Known CHF
* Unstable Angina
* Hb level below 7.5 g/dL or above 8.5 g/dL
* No plan for future transfusion.
* Patient enrollment will happen after patient has consented and scheduled their first/next transfusion.
* Patient will not be enrolled if no future transfusions are scheduled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Abel, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abel GA, Klepin HD, Magnavita ES, Jaung T, Lu W, Shallis RM, Hantel A, Bahl NE, Dellinger-Johnson R, Winer ES, Zeidan AM. Peri-transfusion quality-of-life assessment for patients with myelodysplastic syndromes. Transfusion. 2021 Oct;61(10):2830-2836. doi: 10.1111/trf.16584. Epub 2021 Jul 12. PMID 34251040

RESULTS

PARTICIPANT FLOW:
Groups:
- Peri-Transfusion QOL Assessment: * Participants will be given a study packet containing a paper copy of the QUALMS
  * Study participants will fill out the survey on the day before their first/next pRBC transfusion.
  * Study participants will receive a second paper copy of the QUALMS, along with a stamped envelope addressed to the appropriate site
  * The second assessment will be scored and compared with the first, and both the patient and provider will be sent a report with the results
  Peri-Transfusion QOL Assessment: Participants will undergo a peri-transfusion quality of life assessment (PTQA) using the Quality of Life in Myelodysplasia Scale (QUALMS)
Period: Overall Study
Arm/Group | Peri-Transfusion QOL Assessment
Started | 62
Completed | 38
Not Completed | 24

BASELINE CHARACTERISTICS:
Arm/Group | Peri-Transfusion QOL Assessment
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Transfusion-dependent [Count of Participants; unit: Participants] — Patients with greater than or equal to 1 transfusion scheduled during 8-week period prior to enrollment
  Participants | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Receipt of Second Transfusion
Description: Assessed via medical record review at two months post index transfusion
Time Frame: Two months
Population: Data not collected.
Arm/Group | Peri-Transfusion QOL Assessment
Number analyzed (Participants) | 0

2. Primary Outcome: Median Difference in Units pRBCs (for Those Transfusion-dependent)
Description: Assessed via medical record review at two months post index transfusion. We identified historical matches for 25 patients (21 from Dana-Farber, 1 from Wake Forest, and 3 from Yale) and compared the median number of red cell units in these patients to the PTQA group over 2 months.
Time Frame: Two months
Population: Data not collected.
Arm/Group | Peri-Transfusion QOL Assessment
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Hospitalizations (for Both Transfusion Groups)
Description: Assessed via medical record review at two months post index transfusion
Time Frame: Two months
Population: Data not collected.
Arm/Group | Peri-Transfusion QOL Assessment
Number analyzed (Participants) | 0

4. Primary Outcome: Number of Clinic Visits (for Both Transfusion Groups)
Description: Assessed via medical record review at two months post index transfusion
Time Frame: Two months
Population: Data not collected.
Arm/Group | Peri-Transfusion QOL Assessment
Number analyzed (Participants) | 0

5. Secondary Outcome: PTQA Utilization
Description: Assessed via follow-up survey at 2 months after index transfusion
Time Frame: Two months
Population: Data not collected.
Arm/Group | Peri-Transfusion QOL Assessment
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Patients With Decisional Regret
Description: Assessed via follow-up survey at 2 months after index transfusion. Of the 38 patients who completed PTQA, 6 did not complete the 2-month follow-up survey, and 1 passed away.
Time Frame: Two months
Measure: Count of Participants; unit: Participants
Arm/Group | Peri-Transfusion QOL Assessment
Number analyzed (Participants) | 31
Participants | 3

7. Secondary Outcome: Perceptions of Impact of PTQA on Care
Description: Percentage of patients reporting that PTQA impacted their treatment decisions. Assessed by a binary (yes/no) on the follow-up survey at 2-months after index transfusion.
Time Frame: Two months
Population: Patients who underwent PTQA, were alive and were willing to complete the 2-month follow-up survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Peri-Transfusion QOL Assessment
Number analyzed (Participants) | 31
Participants | 24

8. Secondary Outcome: Perceived Stress by the Associated Scales
Description: Assessed via follow-up survey at 2 months after index transfusion
Time Frame: Two months
Population: Data not collected.
Arm/Group | Peri-Transfusion QOL Assessment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed from baseline (index transfusion) to 1 year.
Description: Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Peri-Transfusion QOL Assessment
All-Cause Mortality (participants affected / at risk) | 1/38
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT03660228/Prot_000.pdf